CLINICAL TRIAL: NCT04952103
Title: Real World Study of Diagnosis and First-line Treatment Among Patients With Cancer of Unknown Primary in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Professor, Fudan University
Other Study IDs: Fudan-CUP-003
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — The patient's treatment is determined by the physician in charge according to the patient's clinical situation and relevant guidelines, without additional intervention.

SUMMARY:
This study is a prospective, real world study.The objective is to observe the diagnosis and first-line treatment of Chinese patients with cancer of unknown primary, and collect the clinicopathological characteristics, treatment outcomes, survival and other data of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Had a diagnosis of cancer of unknown primary (CUP) after a standard evaluation .
* Prepared to receive first-line therapy for CUP

Exclusion Criteria:

* Patients who had previously received systemic therapy for CUP
* Previous history of other cancers, except cervix cancer or basal cell carcinoma of the skin that has been cured
* The investigator considered that there were contraindications to treatment or were not appropriate to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer of unknown primary (CUP) and are gonging to receive the first-line therapy for CUP
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-06-18 (Estimated); Study Completion 2024-06-18 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cencer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided